CLINICAL TRIAL: NCT06067529
Title: A Multicenter Observational Study on the Development and Health Effects of Premature Ovarian Insufficiency
Acronym: POI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhou Jianhong, Department director, Women's Hospital School Of Medicine Zhejiang University
Other Study IDs: ZDFY2022-4XA101
Record Dates: First submitted 2023-07-06; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Premature Ovarian Insufficiency
Keywords: Premature Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premature ovarian insufficiency group
  Interventions: Drug: hormone replacement therapy

INTERVENTIONS:
Drug: hormone replacement therapy — hormone replacement therapy

SUMMARY:
Premature ovarian insufficiency (POI) refers to the occurrence of ovarian hypofunction in women before the age of 40, which seriously affects women's overall health and quality of life. However, there is currently insufficient understanding of the risk factors, pathogenesis, short-term and long-term health effects of POI, and the health effects of the disease, and there is a lack of high-quality evidence to support clinical diagnosis and treatment decisions. This study intends to construct a hospital-based multi-center POI case-control and prospective special disease cohort, after baseline assessment and follow-up monitoring, collect disease characteristics, lifestyle, social psychology, environmental and occupational exposure, biological samples and other data, aiming to observe POI The natural occurrence, progression and health impact of POI, clarify the risk factors of POI, evaluate the impact of POI on women's health and disease risk, and discuss the benefits, risks and options of HRT for POI patients. The results of this study will deepen and expand the understanding of the occurrence and development of POI and its short-term and long-term health effects, provide high-level evidence for optimizing POI prevention, diagnosis and treatment strategies, and establish a long-term management system, laying the foundation for interventional research.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39 years old
* Meet POI diagnostic criteria
* Volunteer to participate in this study and willing to cooperate with the investigation

Exclusion Criteria:

* Reproductive endocrine disease
* Those receiving hormone supplementation and other steroid-containing drug therapy now or within half a year
* Chromosomal abnormalities
* Pregnancy and breastfeeding women
* Uncontrolled endocrine system diseases
* Uncontrolled cardiovascular system diseases
* Uncontrolled autoimmune related diseases
* Abnormal liver function
* Abnormal kidney function
* Abnormal coagulation function
* Severe anemia
* History of malignant tumors
* History of radiotherapy
* History of chemotherapy
* Mental impairment
* Cognitive impairment

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females aged 18-39 who were diagnosed with POI
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
bone density | 1 year
  Dual Energy X-ray
procollagen type I carboxyl-terminal propeptide | 1 year
  peripheral venous blood
fasting blood glucose | 1 year
  peripheral venous blood
Low-density lipoprotein cholesterol/High-density lipoprotein cholesterol | 1 year
  peripheral venous blood
Estradiol/follicle stimulating hormone | 1 year
  peripheral venous blood

SECONDARY OUTCOMES:
free triiodothyronine/free thyroxine | 1 year
  peripheral venous blood

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No